CLINICAL TRIAL: NCT04978870
Title: Diagnosis, Incidence and Consequences of Postoperative Delirium in Elderly Patients in the Post-anaesthetic Care Unit
Brief Title: Diagnosis, Incidence and Consequences of PACU-Delirium
Acronym: PADE-DIC
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-10331-BO-ff
Record Dates: First submitted 2021-06-25; First posted 2021-07-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Delirium; Elderly Patient; Cognitive Decline
Keywords: Post-anesthetic care; Cognitive recovery; Delirium
MeSH Terms: conditions — Emergence Delirium; Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1 - Validation: Group 1 will be screened for delirium during the PACU stay using the CAM-PACU. Delirium criteria as defined by ICD-10 will be assessed in comparison. A subgroup of patients will receive an additional delirium screening using the CAM-PACU. This screening will be performed by another operator blinded for the results from the initial delirium screening.
- 2 - Cognition: Group 2 will be screened for delirium during the PACU stay using the CAM-PACU. Delirium criteria as defined by ICD-10 will be assessed in comparison.
  This group will undergo additional assessment of preoperative and postoperative cognitive function as well as a POD screening using the 3D-CAM starting at postoperative day 1 until discharge from hospital but no longer than postoperative day 5.

SUMMARY:
This study aims to

1. determine sensitivity and specificity of the Confusion Assessment Method for Postanesthesia Care Unit (CAM-PACU)
2. examine the effect of postanesthesia care unit delirium (PACU delirium) on the emergence of later onset postoperative delirium (POD) as well as cognitive recovery until one month postoperatively

ELIGIBILITY:
Inclusion Criteria:

* planned surgery in the near future
* surgery time at least 60min

Exclusion Criteria:

* intracranial surgery
* expected postoperative transfer to ICU and stay exceeding 24h
* length of postoperative stay in hospital below 24h
* insufficient German language skills
* current alcohol or drug misuse
* manifest mental illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients meeting inclusion criteria and presenting for sheduled surgery at the University Medical Centre Hamburg, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Group 1: Sensitivity and specificity of "Confusion Assessment Method - Postanesthetic Care Unit" (CAM-PACU) | 15-240 minutes postoperatively
  in reference to International Classification of Diseases-Version 10 (ICD-10)
Group 2: postoperative delirium after discharge from Postanesthetic Care Unit | 0-5 days postoperatively
  3D CAM and/or medical record

SECONDARY OUTCOMES:
re-test reliability | 15-240 minutes postoperatively
  CAM-PACU
cognitive performance | before, 7 and 30 days postoperatively
  Montreal Cognitive Assessment (MoCA, 0-30 points, higher score = better outcome), Cognitive Telephone Screening Instrument (COGTEL), Patient Reported Outcomes Measurement Information System (PROMIS Neuro QoL)
postoperative complications | 30 days postoperatively
  European Perioperative Clinical Outcome (EPCO) definitions; Standardised Endpoints in Perioperative Medicine - Core Outcome Measures in Perioperative and Anaesthetic Care (Step-COMPAC) definitions
feasibility of delirium screening by questioning of medical staff | before, 3 and 12 months after implementation of CAM-PACU
  self-designed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hamburg University Medical Centre Eppendorf, Hamburg, Hamburg, Germany